CLINICAL TRIAL: NCT06898060
Title: A Multicenter, Randomized, Open-label, Parallel Controlled, Phase III Clinical Study to Evaluate the Efficacy and Safety of Abaloparatide Injection (QLG2128) in the Treatment of Postmenopausal Women With Osteoporosis and at High Risk of Fracture
Brief Title: To Evaluate the Efficacy and Safety of Abaloparatide Injection (QLG2128) in the Treatment of Postmenopausal Women With Osteoporosis and at High Risk of Fracture
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QLG2128-301
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Postmenopausal Women With Osteoporosis
MeSH Terms: interventions — Teriparatide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QLG2128 (Experimental)
  Interventions: Drug: QLG2128
- Teriparatide Injection (Active Comparator)
  Interventions: Drug: Teriparatide Injection

INTERVENTIONS:
Drug: QLG2128 — Recommended dosage is 80 μg subcutaneously once daily，52week
  Arms: QLG2128
Drug: Teriparatide Injection — Recommended dosage is 20μg subcutaneously once daily，52week
  Arms: Teriparatide Injection

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of QLG2128 in the treatment of postmenopausal women with osteoporosis and at high risk of fracture.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women who can walk freely (≥50 and ≤85 years);
* The patient has a body mass index(BMI) of 17.0 kg/m2 to 30 kg/m2；
* The patient has a bone mineral density T-score≤-2.5 and > -5.0 at the lumbar spine (L1-L4) or femoral neck or total hip by dual energy x-ray absorptiometry (DXA)；
* The patient has at least one of the following high risk factors of fracture: 1) history of previous fragility fractures; 2) family history of hip fragility fracture; 3) age≥70 years; 4) BMI≤19.0 kg/m2；5) Currently smoking.
* The patient with at least 2 consecutive vertebrae(L1 to L4) and at least 1 hip can be evaluated for BMD.

Exclusion Criteria:

* In addition to postmenopausal osteoporosis, the other diseases affecting bone metabolism；
* History of osteosarcoma；
* History of orthostatic hypotension；
* Currently suffering from active urinary calculus；
* Received anti-osteoporosis treatment that does not meet protocol requirements；
* Received medication that affects bone metabolism within 4 weeks prior to screening, or is planned to use prohibited drugs/non-drug therapy under the protocol during the study period.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Bone Mineral Density (BMD) of Lumbar Spine From Baseline to 52 Week | Baseline to 52 Week
  Percent Change in Bone Mineral Density (BMD) of Lumbar Spine From Baseline to 52 Week

SECONDARY OUTCOMES:
Percent Change in Bone Mineral Density (BMD) of Lumbar Spine From Baseline to 26 Week | Baseline to 26 Week
  Percent Change in Bone Mineral Density (BMD) of Lumbar Spine From Baseline to 26 Week
Percent Change in Bone Mineral Density (BMD) of Total Hip, Femoral Neck From Baseline to 26/52 Week | Baseline to 26/52 Week
  Percent Change in Bone Mineral Density (BMD) of Total Hip, Femoral Neck From Baseline to 26/52 Week
Proportion of Subjects With New Fragility Fractures From Baseline to 26/52 Week | Baseline to 26/52 Week
  Proportion of Subjects With New Fragility Fractures From Baseline to 26/52 Week